CLINICAL TRIAL: NCT00883675
Title: Multicenter Exploratory Trial of the Safety and Efficacy of Adjuvant Docetaxel and Carboplatin in Patients With Resected Non-small Cell Lung Cancer
Brief Title: Safety Study of Adjuvant Docetaxel-Carboplatin Treatment for Resected Lung Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Mann (Network)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Michael Mann, Director, Maestro Clinical, Inc.
Organization: Maestro Clinical, Inc. (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC#08-002; IIT 12230
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer; Adjuvant therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Docetaxel: 75 mg/m2 over 1 hour every 3 weeks for 3 doses Carboplatin Area Under the Curve 5.5 over 0.5 to 1 hour every 3 weeks for 3 doses
  Interventions: Drug: Docetaxel-Carboplatin

INTERVENTIONS:
Drug: Docetaxel-Carboplatin — Docetaxel: 75 mg/m2 over 1 hour every 3 weeks for 3 doses Carboplatin AUC 5.5 over 0.5 to 1 hour every 3 weeks for 3 doses
  Other Names: Taxotere, Paraplatin

SUMMARY:
The purpose of this study is to determine whether it is safe to treat lung cancer patients who have undergone an attempt at curative resection with the combination of docetaxel and carboplatin.

DETAILED DESCRIPTION:
Patients with stage Ib - IIIa NSCLC participated in an open-label, single arm study to assess the safety and tolerability of docetaxel (75 mg/kg) and carboplatin (AUC 5.5) administered for 3 cycles after resection for curative intent. The primary endpoint of the study was safety, as reflected by a febrile neutropenia rate of <10%. Other endpoints assessed protocol compliance and the impact of minimally invasive surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer stage IB - IIIA, complete resection with mediastinal lymph node dissection
* ECOG status 0-1
* >14 and <56 days since resection

Exclusion Criteria:

* Prior chemotherapy and/or radiation therapy for lung cancer
* Peripheral neuropathy > grade 1
* Concurrent other malignancies, other than basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Medical condition that will not permit treatment or follow up according to the protocol
* Prior treatment with docetaxel or carboplatin
* Hypersensitivity to polysorbate 80, platinum-containing compounds or mannitol
* Treatment with other investigational anti-cancer drugs within 30 days of registration
* Pregnant or nursing women
* HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jablons, MD, Principal Investigator — Maestro Clinical
Locations (12):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States
- China (11):
  - Beijing Chaoyang Hospital, Beijing
  - Beijing Tumor Hospital, Beijing
  - Beijing Youyi Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Xuanwu Hospital, Beijing
  - First Affiliated Hospital, Guangzhou Medical College, Guangzhou
  - Sun Yat-sen Cancer Center, Guangzhou
  - Shanghai Chest Hopsital, Pulmonary Medicine, Shanghai
  - Shanghai Lung Cancer Center, Shanghai Chest Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Tianjin Cancer Center, Tianjin

REFERENCES:
- [Derived] Zhi X, Gao W, Han B, Yang Y, Li H, Liu D, Wang C, Min G, Long H, Rigas JR, Carey M, Jahan T, Sammann A, Reza J, Wang D, Mann MJ, Jablons DM, He J; China Clinical Trials Consortium. VATS lobectomy facilitates the delivery of adjuvant docetaxel-carboplatin chemotherapy in patients with non-small cell lung cancer. J Thorac Dis. 2013 Oct;5(5):578-84. doi: 10.3978/j.issn.2072-1439.2012.02.05. PMID 24255769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of patients took place at a single center in the United States (Dartmouth-Hitchcock Norris Cotton Cancer Center) and at ten sites in China that were early members of the China Clinical Trials Consortium.
Period: Overall Study
Arm/Group | Treatment
Started | 133
Completed | 133
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Docetaxel: 75 mg/m2 over 1 hour every 3 weeks for 3 doses Carboplatin Area Under the Curve (AUC) 5.5 over 0.5 to 1 hour every 3 weeks for 3 doses
Arm/Group | Treatment
Number analyzed (Participants) | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 87
  >=65 years | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 59.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 89
Region of Enrollment [Number; unit: participants]
  United States | 2
  China | 131

OUTCOME MEASURES:

1. Primary Outcome: Febrile Neutropenia
Description: The primary endpoint of the study was safety, as reflected by a febrile neutropenia rate of <10%.
Time Frame: 2 months
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 133
participants | 12

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 14/133
Other Adverse Events (participants affected / at risk) | 66/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=133)
Allergic Reaction (Immune system disorders) | 4 (4) — 4 allergic reactions to docetaxel that required discontinuation of therapy
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Infection (Blood and lymphatic system disorders) | 3 (3)
Severe Neutropenia (Blood and lymphatic system disorders) | 3 (4) — requiring hospitalization
Severe Nausea and Vomiting (Gastrointestinal disorders) | 2 (4) — Requiring Hospitalization
Pelvic Infection (Infections and infestations) | 1 (1) — Requiring Hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=133)
Febrile Neutropenia (Infections and infestations) | 11 (11) — Resolved without serious complication
Neutropenia (Blood and lymphatic system disorders) | 55 (55) — Grade 3 and Grade 4 Neutropenia, non-febrile

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days